CLINICAL TRIAL: NCT02115035
Title: A Phase II Single Agent Study to Evaluate the Overall Response Rate, Safety and Tolerability of Orally Administered Vemurafenib (VMRB) in Patients With Relapsed or Refractory Multiple Myeloma Who Have Activated BRAF Mutation
Brief Title: A Single Agent Study to Evaluate the Overall Response Rate, Safety and Tolerability of Orally Administered Vemurafenib
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding issues
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vermurafenib (Experimental): Vermurafenib dosing will be given twice daily by oral administration in cycles of 28 days
  Interventions: Drug: Vermurafenib

INTERVENTIONS:
Drug: Vermurafenib — 960 mg of Vermurafenib twice daily orally on a 28 day schedule
  Other Names: RO5185426; PLX4032

SUMMARY:
The objective is to evaluate the overall response rate of Vermurafenib when administered orally to patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is an open-label study to evaluate the objective response rates of orally administered Vermurafenib for patients with double refractory multiple myeloma. Double refractory multiple myeloma is myeloma that has become refractory to two chemotherapeutic agents such as bortexomib and lenalidomide. The study will be conducted in two stages with an interim data analysis performed after enrollment of the initial 21 subjects to determine whether the study will enroll an additional 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Been identified as having multiple myeloma with activating NRAS, KRAS or BRAF genetic mutations on CD138+ cells, identified by F1 testing
* Have been diagnosed with multiple myeloma by having met all three of the following IMWG criteria:
* Clonal bone marrow plasma cells >10%
* Presence of serum and/or urinary M-protein
* Evidence of end-organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically, one or more of the following:

  * Hypercalcemia: serum calcium >11.5 mg/100 mL
  * Renal insufficiency: serum creatinine >2 mg/dL
  * Anemia: normochromic, normocytic with a hemoglobin value >2 g/100 mL below the lower limit of normal or a hemoglobin value <10 g/100 mL
  * Bone lesions: lytic lesions, severe osteopenia, or pathologic fractures
* Have measurable disease defined by the following:
* Serum M-protein ≥1g/dL or urine M-protein ≥200 mg/24 hours by protein electrophoresis
* If neither serum nor urine M-protein meet the criteria above, then kappa or lambda serum FLC must be ≥10 mg/dL accompanied by an abnormal kappa to lambda ratio (<0.26 or >1.65) (Serum FLC should only be used for patients without measurable serum or urine M-protein spike.)
* Have relapsed or refractory disease after two or more prior multiple myeloma treatment regimens, each of which may have consisted of either single or multiple therapies
* Patient must be at least 3 weeks beyond the last multiple myeloma therapy and any previous therapy related toxicities must be CTCAE (Version 3.0) ≤ Grade 2 (except alopecia)
* Have an Zubrod Performance Status of 0 to 2 (Appendix D)
* Have life expectancy of at least 3 months in the opinion of the enrolling investigator
* Be ≥18 years of age and willing to provide written informed consent
* For women and men of childbearing potential, must have used effective contraceptive methods for previous 4 weeks and agree to continue using such methods during the study and for at least 4 weeks after completing the study, this must include two forms of birth control, including surgical sterilization, a reliable barrier method with spermicide, birth control pills, or contraceptive hormone implants.
* Women of childbearing potential must have a negative serum pregnancy test within 24 hours before the initiation of VMFB therapy.
* Have an absolute neutrophil count >1,000/mm3
* Unsupported platelet count >35,000/mm3
* Have total direct bilirubin <2.0 mg/dL
* Have aspartate aminotransferase and alanine aminotransferase ≤3 times the upper limit of normal
* Have serum Creatinine ≤2.5 times the upper limit of normal
* Have hemoglobin ≥8.5 g/dL
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels

Exclusion Criteria:

* Have non-secretory myeloma
* Have evaluable disease only according to CRAB diagnostic criteria and International Staging System (ISS)
* No previous history of NRAS/KRAS/BRAF inhibitor
* Have an active infection or ,in the opinion of the enrolling investigator, have a serious comorbid medical condition
* Be receiving other concurrent anticancer agents or therapies
* Be receiving other concurrent investigational therapies or have received investigational therapies within 3 weeks of enrollment
* In the opinion of the enrolling investigator, be eligible to receive any other standard therapy available that is known to extend life expectancy
* Be pregnant, nursing, unwilling or unable to utilize two forms of birth control, including surgical sterilization, a reliable barrier method with spermicide, birth control pills, or contraceptive hormone implants.
* Have a history of another malignancy, except as noted below Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer and/or subjects with indolent second malignancies are eligible.
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures as determined by the enrolling investigator
* History of interstitial lung disease or pneumonitis.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to study drug, or excipients or to dimethyl sulfoxide (DMSO).
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrollment.
* Current use of a prohibited medication (Appendix F).
* History of retinal vein occlusion (RVO)
* Symptomatic or untreated spinal cord compression.
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).
* History cardiovascular risk including any of the following:

  * Ejection fraction by ECHO or MUGA must be > 40% and must be performed within 60 days prior to enrollment, unless the patient has received chemotherapy within that period of time in which case the LVEF must be repeated
  * New York Heart Association (NYHA) Class III or Class IV heart failure
  * History or evidence of current clinically significant uncontrolled arrhythmias. NOTE: Exception: Subjects with controlled atrial fibrillation for >30 days prior to study enrollment
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study enrollment
  * Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy;
  * Patients with intra-cardiac defibrillators;
  * Known cardiac metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Changes in serum values | 3 year
  To determine the changes in serum values of monoclonal protein

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh Jethava, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States